CLINICAL TRIAL: NCT05656001
Title: Examining the Effects of Real-time fMRI Neurofeedback and Biofeedback in Adolescents With Nonsuicidal Self-injury
Brief Title: Neuro- and Biofeedback in Nonsuicidal Self-injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Maria Zetterqvist, Principal investigator, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-04702
Record Dates: First submitted 2022-01-31; First posted 2022-12-19 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Nonsuicidal Self Injury; Emotion Regulation
Keywords: nonsuicidal self-injury; emotion regulation; adolescents; neurofeedback; biofeedback
MeSH Terms: conditions — Self-Injurious Behavior; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either an active feedback intervention or a control condition, consisting of a sham feedback.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the outcomes assessor will not know if the participants receive actual or sham feedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real-time functional magnetic resonance imaging neurofeedback and real-time biofeedback (Experimental): Three sessions of real-time functional magnetic resonance imaging neurofeedback (rt-fMRI-NF) or real-time biofeedback training where participants will receive direct visual feedback from the blood oxygenation level dependent (BOLD) imaging signaling from the salience network in rt-fMRI-NF or visual feeback from a physiological signal in the real-time biofeedback (active condition)
  Interventions: Other: Real-time functional magnetic resonance imaging Neurofeedback and Real-time Biofeedback
- Sham feedback (Sham Comparator): Three session where participants will be given a yoked sham feedback as control condition.
  Interventions: Other: Sham functional magnetic resonance imaging neurofeedback and sham biofeedback

INTERVENTIONS:
Other: Real-time functional magnetic resonance imaging Neurofeedback and Real-time Biofeedback — Participants will take part in three runs of real-time functional magnetic resonance imaging feedback (rt-fMRI-NF) training with 4-8 days apart, which will be conducted at the Center for Medical Image Science and Visualization (CMIV) at the university hospital in Linköping. Participants who receive biofeedback will take part in three runs of biofeedback with 4-8 days apart conducted in the lab at the Center for Social and Affective Neuroscience (CSAN) at Linköping university. Participants will be given instructions and basic psychoeducation of brain function and the rational for down-regulating the area of the brain that drives emotion, as well as the physiological reaction that is triggered in response to emotional stimuli. The emotional stimuli are emotional pictures from the International Affective Picture System (IAPS) and the Open Affective Standardized Image Set (OASIS).
  Arms: real-time functional magnetic resonance imaging neurofeedback and real-time biofeedback
Other: Sham functional magnetic resonance imaging neurofeedback and sham biofeedback — Participants will take part in three runs of sham neurofeedback with 4-8 days apart, which will be conducted at the Center for Medical Image Science and Visualization (CMIV) at the university hospital in Linköping. Participants who receive sham biofeedback will take part in three runs of sham biofeedback with 4-8 days apart conducted in the lab at the Center for Social and Affective Neuroscience (CSAN) at Linköping university. Participants will be given instructions and basic psychoeducation of brain function and the rational for down-regulating the area of the brain that drives emotion, as well as the physiological reaction that is triggered in response to emotional stimuli. The emotional stimuli are emotional pictures from the International Affective Picture System (IAPS) and the Open Affective Standardized Image Set (OASIS).
  Arms: Sham feedback

SUMMARY:
Nonsuicidal self-injury (NSSI) is defined as the direct, deliberate destruction of one's own body tissue without suicidal intent, typically including behaviors such as cutting, burning, or hitting oneself. The risk of engaging in NSSI is particularly high during adolescence. NSSI is associated with impairments in emotion regulation and NSSI behavior serves as an attempt to regulate emotion. We propose to examine whether training adolescents with NSSI to self-regulate using emotion regulation skills to down-regulate hemodynamic activity of the salience network, involved in emotional processing. Moreover, we propose to examine whether limbic-prefrontal cortex connectivity can be increased following neurofeedback, thereby helping adolescents find an optimal way to emotionally regulate with the help of neurofeedback, instead of engaging in NSSI to regulate emotions. We also aim to examine effects of real-time biofeedback by investigating if adolescents can regulate their psychophysiological activity during emotional reactivity with biofeedback. Sixty participants with NSSI will be recruited and offered either real-time functional magnetic resonance imaging (rt-fMRI-NF) (n = 30) or real-time biofeedback (n = 30) training. Participants each each condition will then be randomized to either an active or a control condition (n = 15/group). Participants will take part in three runs of feedback training. Changes in emotional reactivity as measured with facial electromyography (EMG) before and after feedback training will be the proximal outcome measure together with changes of the blood oxygenation level dependent (BOLD) response during real-time fMRI-neurofeedback for the neurofeedback training. Proximal outcome measures for the biofeedback will include psychophysiological measures of emotional reactivity (facialEMG). More distal outcome measures for both neuro- and biofeedback will be measures of NSSI: frequency, methods and severity as well as self-report measures of difficulties with regulating emotions, emotional reactivity and psychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* ongoing contact at the child- and adolescent psychiatric clinics in both Linköping and Norrköping, Sweden
* ongoing contact at the primary care facilities in Linköping and Norrköping (Ungdomshälsan, Råd, Stöd & Hälsa)
* NSSI, independent of psychiatric diagnosis
* between 15 and 19 years of age
* having engaged in five or more instances of NSSI during the last six months
* the patient is cognitively capable to decide for him- or herself

Exclusion Criteria:

* anorexia in starvation with BMI 16 or under
* substance abuse disorder
* psychosis
* needing interpreter
* intellectual disability
* and for those who do the neurofeedback, severe claustrophobia, pregnancy and braces

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Emotional reactivity | Change from baseline up to 5 weeks
  Changes of emotional reactivity is measured with facial electromyography (facialEMG). High zygomatic and corrugator response indicate higher emotional reactivity.
Hemodynamic activity | Change from baseline at up to 4 weeks
  Changes of the blood oxygenation level dependent (BOLD) response during real-time fMRI-neurofeedback for the neurofeedback training. The aim is to down-regulate the hemodynamic activity in the salience network.
Psychophysiological response | Change from baseline at up to 4 weeks
  Changes of psychophysiological response during the real-time biofeedback training. The aim is to decrease the emotional reactivity and psychophysiological response.

SECONDARY OUTCOMES:
Nonsuicidal self-injury | Change from baseline at up to 5 weeks, and at additional 6 weeks and 3 month follow-up
  Changes of self-reported frequency in nonsuicidal self-injury (NSSI). NSSI frequency is measured using the short 9-item version of the Deliberate Self-Harm Inventory (DSHI). Open ended questions are used for frequency with a range from 0 to several hundreds, depending on participants answers. Higher scores indicate more NSSI frequency and worse outcome.
Difficulties with emotion regulation | Change from baseline at up to 5 weeks, and at additional 6 weeks and 3 month follow-up
  Changes of self-reported difficulties with emotion regulation. Difficulties with emotion regulation is measured using the 16-item version of the Difficulties with Emotion Regulation Scale (DERS-16). Scores range from 16 to 80 where higher scores indicate more difficulties with emotion regulation.
Emotional reactivity | Change from baseline at up to 5 weeks, and at additional 6 weeks and 3 month follow-up
  Changes of self-reported emotional reactivity. Emotional reactivity is measured with the Emotion Reactivity Scale (ERS). Total scores range from 0 to 84 and a higher score indicates a worse outcome.
Emotional awareness | Change from baseline at up to 5 weeks, and at additional 6 weeks and 3 month follow-up
  Changes of self-reported emotional awareness. Emotional awareness is measured with Toronto Alexithymia Scale, 20 items (TAS-20). TAS-20 total score ranges from 20 to 100 and higher scores indicate worse outcome.
Psychiatric symptoms | Change from baseline at up to 5 weeks, and at additional 6 weeks and 3 month follow-up
  Changes of self-reported psychiatric symptoms. Psychiatric symptomatology is measured with the Trauma Symptom Checklist for Children (TSCC) with subscales: depression, anxiety, dissociation, posttraumatic stress, anger and sexual preoccupation. The total scale ranges from 0 to 162 and higher scores indicate worse outcome.
Self-criticism | Change from baseline at up to 5 weeks, and at additional 6 weeks and 3 month follow-up
  Changes of self-reported levels of self-criticism. Self-criticism is measured with the Self-Rating Scale (SRS). Scores range from 8 to 56, and higher scores indicate higher levels of self-criticism.
Functions of nonsuicidal self-injury | Change from baseline at up to 5 weeks, and at additional 6 weeks and 3 month follow-up
  Changes of self-reported levels of nonsuicidal self-injury (NSSI) functions. NSSI functions is measured using Clinical Assessment of Nonsuicidal Self-Injury Disorder Index (CANDI). Functions are rated as percentages and scores range from 0 to 100% where higher scores indicate higher usage of a specific NSSI function.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Zetterqvist, PhD, Principal Investigator — Region Östergötland and Linköping university
Locations (1):
- Region Östergötland, Linköping, Sweden